CLINICAL TRIAL: NCT02580058
Title: A PHASE 3, MULTICENTER, RANDOMIZED, OPEN-LABEL STUDY OF AVELUMAB (MSB0010718C) ALONE OR IN COMBINATION WITH PEGYLATED LIPOSOMAL DOXORUBICIN VERSUS PEGYLATED LIPOSOMAL DOXORUBICIN ALONE IN PATIENTS WITH PLATINUM-RESISTANT/REFRACTORY OVARIAN CANCER
Brief Title: A Study Of Avelumab Alone Or In Combination With Pegylated Liposomal Doxorubicin Versus Pegylated Liposomal Doxorubicin Alone In Patients With Platinum Resistant/Refractory Ovarian Cancer (JAVELIN Ovarian 200)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991009; 2015-003091-77 (EudraCT Number); JAVELIN OVARIAN 200 (Other: Alias Study Number)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer
Keywords: platinum resistant; platinum refractory
MeSH Terms: conditions — Ovarian Neoplasms | interventions — avelumab; 1-dodecylpyridoxal; Doxorubicin; liposomal doxorubicin

ARMS (3):
- avelumab (Experimental): Arm A: avelumab alone
  Interventions: Biological: avelumab
- avelumab plus pegylated liposomal doxorubicin (PLD) (Experimental): Arm B: avelumab plus PLD
  Interventions: Biological: avelumab; Drug: PLD
- PLD (Active Comparator): Arm C: PLD alone
  Interventions: Drug: PLD

INTERVENTIONS:
Biological: avelumab — 10 mg/kg will be given as a 1 hour intravenous infusion (IV) every 2 weeks (Q2W) in 4 week cycles
  Arms: avelumab; avelumab plus pegylated liposomal doxorubicin (PLD)
Drug: PLD — PLD (Arm B, Arm C) 40 mg/m2 will be given as a 1 hour IV infusion every 4 weeks (Q4W) in 4 week cycles
  Other Names: doxorubicin, caelyx
  Arms: PLD; avelumab plus pegylated liposomal doxorubicin (PLD)

SUMMARY:
A Phase 3 global study comparing avelumab alone to avelumab plus PLD and to PLD alone to demonstrate that avelumab given alone or in combination with PLD is superior to PLD alone in prolonging Overall Survival in patients with platinum resistant/platinum refractory ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian, fallopian tube, or peritoneal cancer, including malignant mixed Müllerian tumors with high grade serous component.
* Platinum resistant/refractory disease, defined as disease progression within 180 days following the last administered dose of platinum therapy (resistant), or lack of response or disease progression while receiving the most recent platinum based therapy (refractory), respectively.
* Received up to 3 lines of systemic anticancer therapy for platinum sensitive disease, most recently platinum containing, and no prior systemic therapy for platinum resistant disease
* Measurable disease by investigator assessment with at least 1 unidimensional measurable lesion by RECIST v.1.1 that has not previously been irradiated
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Patients with diabetes type I, vitiligo, psoriasis, hypo or hyperthyroid disease not requiring immunosuppressive treatment are eligible.

Mandatory tumor biopsy must be performed prior to enrollment for all patients (unless there is a documented clinical contraindication). In addition, availability of archived FFPE tumor tissue should be confirmed. If a patient underwent tumor tissue collection within 3 months prior to enrollment with no intervening treatment, and the sample is provided, then a new de novo tumor biopsy is not required.

Exclusion Criteria:

* Non epithelial tumor or ovarian tumors with low malignant potential (ie, borderline tumors).
* Prior therapy with an anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti cytotoxic T lymphocyte associated antigen 4 (CTLA 4) antibody (including ipilimumab, tremelimumab or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways).
* Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 4 weeks prior to study entry and are neurologically stable.
* Diagnosis of any other malignancy within 5 years prior to registration, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix.
* Severe gastrointestinal conditions such as clinical or radiological evidence of bowel obstruction within 4 weeks prior to study entry, uncontrolled diarrhea in the last 4 weeks prior to enrollment, or history of inflammatory bowel disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 566 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (284):
- United States (80):
  - Arizona Oncology Associates, PC - HAL, Chandler, Arizona
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Scottsdale, Arizona
  - Arizona Oncology Associates, PC-HAL, Tempe, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - University of California, Irvine/UC Irvine Health, Orange, California
  - Sansum Clinic, Santa Barbara, California
  - Sansum Clinic, Solvang, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Florida Cancer Specialists, Daytona Beach, Florida
  - Florida Cancer Specialists, Wellington, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Atlanta Gynecologic Oncology, Atlanta, Georgia
  - Northside Hospital - Pharmacy, Atlanta, Georgia
  - University Gynecologic Oncology, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, P.C., Austell, Georgia
  - Northwest Georgia Oncology Centers, P.C., Carrollton, Georgia
  - Northwest Georgia Oncology Centers, P.C., Cartersville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Douglasville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Norton Healthcare Pharmacy, Attn: Marlon Baranda, Pharm D, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - Maryland Oncology Hematology, P.A., Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Maryland Oncology Hematology P.A., Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The University of Kansas Cancer Center, CCP - North, Kansas City, Missouri
  - Center of Hope at Renown Regional Medical Center, Reno, Nevada
  - Southwest GYN Oncology Associates, Inc., Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - Mission Hospital, Inc., Asheville, North Carolina
  - Novant Health Oncology Specialists, Kernersville, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Fairview Hospital Moll Pavilion Cancer Center, Cleveland, Ohio
  - Fairview Hospital Moll Pavilion Pharmacy, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hillcrest Hospital Hirsch Cancer Center Pharmacy, Mayfield Heights, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Investigational Drug Services, University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology-South Austin, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology -Fort Worth Cancer Center, Fort Worth, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center, Irving, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Carilion Clinic Gynecologic Oncology, Roanoke, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (19):
  - Epic Pharmacy,Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Newcastle Private Hospital Pty Limited, Newcastle, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Rivercity Pharmacy, Auchenflower, Queensland
  - Mater Pharmacy Services, Brisbane, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Clinical Research Unit, Herston, Queensland
  - Metro North Hospital and Health Service, Herston, Queensland
  - Oncology Pharmacy, Herston, Queensland
  - Icon Cancer Care, South Brisbane, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Cabrini Health Limited, Brighton, Victoria
  - Cabrini Health Limited, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Pharmacy Department, Parkville, Victoria
  - The Royal Women's Hospital, Parkville, Victoria
- Austria (2):
  - Medizinische Universitat Graz, LKH-Univ. Klinikum Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
- Belgium (6):
  - University Hospital Gent, Ghent, EAST Flanders
  - Institut Jules Bordet, Brussels
  - AZ Groeninge Hospital, Kortrijk
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHU de Liege - Sart Tilman, Liège
  - Clinique et Maternite Sainte Elisabeth, Namur
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Sindi Ahluwalia Hawkins Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency-Vancouver Centre, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Health Authority, QEII Health Sciences Centre, Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Nova Scotia Health Authority, QEII Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - Oncology Pharmacy McGill University Health Centre, Montreal, Quebec
- Czechia (8):
  - Vseobecna fakultni nemocnice v Praze, Fakultni poliklinika, Prague, Czech Republic
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice v Praze, Nemocnicni lekarna,, Prague
  - Vseobecna fakultni nemocnice v Praze, Neurologicka klinika, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
  - Krajska zdravotni a.s., Masarykova nemocnice v Usti nad Labem, o.z, Ústí nad Labem
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
- France (8):
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Service de Radiologie, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus, Villejuif
- Greece (2):
  - General Hospital of Athens Alexandra, Athens
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", 2nd Department of Medical Oncology, Athens/New Kifissia
- Hong Kong (2):
  - Princess Margaret Hospital, Hong Kong
  - University of Hong Kong, Hong Kong
- Hungary (5):
  - Orszagos Onkologiai Intezet, Gyogyszertar, Budapest
  - Orszagos Onkologiai Intezet, Nogyogyaszati Osztaly, Budapest
  - Debreceni Egyetem Klinikai Gyogyszertar, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Onkologiai Kozpont, Szolnok
- Ireland (8):
  - Mater Misericordiae University Hospital, Dublin, Dublin
  - Mater Private Hospital, Dublin, Dublin
  - St James's Hospital, Dublin
  - Mater Misericoridae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - Pharmacy Department, Dublin
  - St Vincent's University Hospital, Dublin
  - University Hospital Waterford, Waterford
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (20):
  - Poliambulatorio Specialistico Villa Salute, Manerbio, Brescia
  - Congregazione delle Suore Infermiere dell'Addolorata, Costa Masnaga, Lecco
  - ASST Fatebenefratelli Sacco, Miano, Milano
  - Servizio Sanitario Regionale Emilia-Romagna, Lugo, Ravenna
  - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Habilita, San Marco Bergamo, Bergamo
  - Humanitas Cliniche Gavazzeni, Bergamo
  - Humanitas, Unita Operativa di Cardiologia 2, Bergamo
  - Fondazione Poliambulanza Istituto Ospedelario, Brescia
  - Congregazione delle Suore Infermiere dell'Addolorata, Como
  - Fondazione Teresa Camplani, Cremona
  - Regione Lombardia, A O Istituti Ospitalieri di Cremona, Cremona
  - Regione Lombardia, ASST Cremona, Cremona
  - Istituto Europeo di Oncologia, Milan
  - Ambulatorio dott. Francesco Cavanna, Medico Chirurgo, Piacenza
  - Azienda Unita Sanitaria Locale di Piacenza, Piacenza
  - Azienda USL 4 Prato, Prato
  - Azienda USL 4 Toscana Centro, Prato
  - Servizio Sanitario Regionale Emilia-Romagna, Rimini
  - C D C, Sede di Torino Centro, Torino
- Japan (19):
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Tokai University Hospital, Isehara, Kanagawa
  - Nippon Medical School Musashikosugi Hospital, Kawasaki, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - National Defense Medical College Hospital, Tokorozawa, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kagoshima University Hospital, Kagoshima
  - Kagoshima City Hospital, Kagoshima
  - Niigata Cancer Center Hospital, Niigata
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - LUMC, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
- Norway (4):
  - Department of Obstetrics and Gynecology, Haukeland University Hospital, Bergen
  - Sykehusapoteket i Bergen, Bergen
  - Oslo Universitetssykehus, Oslo
  - Sykehusapoteket Oslo, Oslo
- Poland (8):
  - Centrum Onkologii, Instytut im. M. Sklodowskiej-Curie, Oddzial w Krakowie, Apteka Szpitalna, Krakow
  - Centrum Onkologii, Instytut im. M. Sklodowskiej-Curie, Oddzial w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Apteka Szpitalna, Olsztyn
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w, Poznan
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego, Poznan
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3 w Rybniku, Apteka Szpitalna, Rybnik
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3 w Rybniku, Rybnik
- Russia (10):
  - State Budgetary Healthcare Institution "Oncology Center #2" of the Ministry of Healthcare, Sochi, Krasnodarskiy Kray
  - State Budgetary Healthcare Institution Pyatigorsk Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - Evimed Llc, Chelyabinsk
  - State Budgetary Healthcare Institution, Chelyabinsk
  - State Budgetary Healthcare Institution "Clinical oncology dispensary #1", Krasnodar
  - Federal State Budgetary Institution "Russian Cancer Research Center n.a. N.N. Blokhin", Moscow
  - State Budgetary Healthcare Institution of Nizhegorogsky region, Nizhny Novgorod
  - State Budgetary Healthcare Institution "Orenburg Regional Clinical Oncological Dispensary", Orenburg
  - State Budget Institution of Healthcare Saint Petersburg Clinical Scientific - Practice Center, Saint Petersburg
  - State Regional Budgetary Healthcare Institution "Regional clinical oncology dispensary", Veliky Novgorod
- Singapore (4):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore Pharmacy, Singapore
  - National Cancer Centre Singapore, Singapore
  - Raffles Hospital, Singapore
- South Korea (13):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Clinical Trial Pharmacy, Keimyung University Dongsan Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Clinical Trial Pharmacy, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center Clinical Trial Pharmacy, Seoul
  - Samsung Medical Center, Seoul
  - Department of Pharamacy, The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul
- Spain (7):
  - Institut Catala d'Oncologia - Hospital Duran y Reynalds, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - lnstitut Catala d Oncologia de Girona. Hospital Universitario Dr. Josep Trueta, Girona
  - Hospital MD Anderson, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Virgen de Valme, Seville
- Switzerland (9):
  - Universitatsspital Basel, Frauenklinik, Basel, Canton of Basel-City
  - Universitatsspital Basel, Basel, Canton of Basel-City
  - Luzerner Kantonsspital, Medizinische Onkologie, Studienzentrale Onkologie, Lucerne, Canton of Lucerne
  - Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Canton Ticino
  - Kantonsapotheke Zurich, Zurich
  - Universitaetsspital Zurich, Klinik fuer Gynakologie, Zurich
  - Universitatsspital Zurich, Clinical Trials Center, Zurich
  - Universitatsspital Zurich, Institut fur diagnostische und interventionelle Radiologie, Zurich
  - Universitatsspital Zurich, Universitares Herzzentrum Zurich, Zurich
- Taiwan (11):
  - Clinical Trial Pharmacy, National Cheng Kung University Hospital, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Clinical Trial Pharmacy, Mackay Memorial Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Clinical Trial Pharmacy, Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Clinical Trial Pharmacy, Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan
  - Chemotherapy Pharmacy, Chang Gung Memorial Hospital - Linkou Branch, Taoyuan
- United Kingdom (18):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Ross Hall Hospital, Glasgow, CITY of Glasgow
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral, Merseyside
  - The Clatterbridge Cancer Centre, Bebington, Wirral, Merseyside
  - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - Northampton General Hospital NHS Trust, Northampton, Northamptonshire
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Spire Healthcare Limited (St. Anthony's Hospital), Sutton, Surrey
  - NHS Greater Glasgow and Clyde, Glasgow
  - University College London Hospital NHS Foundation Trust, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Guy's & St. Thomas' NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie Hospital NHS Foundation Trust, Manchester
  - Nottingham University Hospital NHS Trust, Nottingham
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bonaca MP, Moslehi JJ, Ledermann JA, Michelon E, Wei C, Moran M, Monk BJ, Pujade-Lauraine E. Left Ventricular Ejection Fraction in Patients With Ovarian Cancer Treated With Avelumab, Pegylated Liposomal Doxorubicin, or Both. Oncologist. 2023 Oct 3;28(10):e977-e980. doi: 10.1093/oncolo/oyad213. PMID 37665777
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Pujade-Lauraine E, Fujiwara K, Ledermann JA, Oza AM, Kristeleit R, Ray-Coquard IL, Richardson GE, Sessa C, Yonemori K, Banerjee S, Leary A, Tinker AV, Jung KH, Madry R, Park SY, Anderson CK, Zohren F, Stewart RA, Wei C, Dychter SS, Monk BJ. Avelumab alone or in combination with chemotherapy versus chemotherapy alone in platinum-resistant or platinum-refractory ovarian cancer (JAVELIN Ovarian 200): an open-label, three-arm, randomised, phase 3 study. Lancet Oncol. 2021 Jul;22(7):1034-1046. doi: 10.1016/S1470-2045(21)00216-3. Epub 2021 Jun 15. PMID 34143970
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B9991009&StudyName=A%20Phase%203%2C%20Multicenter%2C%20Randomized%2C%20Open-label%20Study%20Of%20Avelumab%20%28msb0010718c%29%20Alone%20Or%20In%20Combination%20With%20Pegylated%20Liposomal%20Doxorubicin%20Versus%20Pegylated%20Liposomal%20Doxorubicin%20Alone%20In%20Patients%20With%20Platinum-resistant%2Frefractory%20Ovarian%20Cancer
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B9991009&StudyName=A+Phase+3%2C+Multicenter%2C+Randomized%2C+Open-label+Study+Of+Avelumab+%28msb0010718c%29+Alone+Or+In+Combination+With+Pegylated+Liposomal+Doxorubicin+Versus+Pegylated+Liposomal+Doxorubicin+Alone+In+Patients+With+Platinum-resistant%2Frefractory+Ovarian+Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data reported based on last participant last visit (LPLV) date (12 July 2022).
Groups:
- Avelumab: Avelumab 10 milligram (mg)/kilogram (kg) given as a 1-hour intravenous (IV) infusion every 2 weeks (Q2W) in 4-week cycles.
- Avelumab + PLD: Avelumab 10 mg/kg given as a 1-hour IV Q2W in 4-week cycles + pegylated liposomal doxorubicin (PLD) 40 mg/square meter given as a 1-hour IV infusion every 4 weeks (Q4W) in 4-week cycles.
- Pegylated Liposomal Doxorubicin (PLD): PLD 40 mg/square meter given as a 1-hour IV infusion Q4W in 4-week cycles.
Period: Overall Study
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Started (This table included all randomized participants.) | 188 | 188 | 190
Treated (Participants received at least 1 dose of study drug.) | 187 | 182 | 177
Completed (Participants were considered completed when at least one drug of the combination is completed.) | 0 | 0 | 0
Not Completed | 188 | 188 | 190
Not completed — Adverse Event | 16 | 30 | 20
Not completed — Death | 4 | 4 | 5
Not completed — Physician Decision | 1 | 3 | 11
Not completed — Other | 5 | 1 | 3
Not completed — Withdrawal by Subject | 4 | 7 | 31
Not completed — Global Deterioration of Health Status | 19 | 18 | 24
Not completed — No Longer Meets Eligibility Criteria | 1 | 0 | 2
Not completed — Progressive Disease | 137 | 125 | 94
Not completed — Non-Compliance With Study Drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD) | Total
Number analyzed (Participants) | 188 | 188 | 190 | 566
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 124 | 114 | 349
  >=65 years | 77 | 64 | 76 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (10.26) | 59.5 (10.05) | 60.4 (10.64) | 60.3 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 188 | 190 | 566
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 176 | 176 | 183 | 535
  Unknown or Not Reported | 10 | 9 | 6 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 2 | 2 | 6 | 10
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 1
  Race: Asian | 34 | 53 | 46 | 133
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Race: White | 148 | 133 | 135 | 416
  Race: Other | 1 | 0 | 2 | 3
  Race: Unknown | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death due to any cause. OS time was summarized by treatment arm using the Kaplan-Meier method.
Time Frame: From randomization until the date of first documented progression or date of deaths from any cause, whichever came first, assessed up to 30 months (based on cutoff date: 19 September 2018).
Population: The primary analyses of OS were performed based on the Full Analysis Set (FAS). The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
months | 11.8 [8.9 to 14.1] | 15.7 [12.7 to 18.7] | 13.1 [11.8 to 15.5]
Statistical Analysis 1: Comparison: Avelumab vs Pegylated Liposomal Doxorubicin (PLD); Test type: Superiority; p = 0.8253, Log Rank; 1-sided; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.867 to 1.497]
Statistical Analysis 2: Comparison: Avelumab + PLD vs Pegylated Liposomal Doxorubicin (PLD); Test type: Superiority; p = 0.2082, Log Rank; 1-sided; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.672 to 1.179]

2. Primary Outcome: Progression Free Survival (PFS) Based on Blinded Independent Central Review (BICR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS is defined as the time from date of randomization to the date of the first documentation of progression of disease (PD) or death due to any cause, whichever occurs first. PFS time was summarized by treatment arm using the Kaplan-Meier method. PFS based on BICR assessment was evaluated for this endpoint.
Time Frame: From randomization to date of first documentation of PD or death due to any cause whichever was first (up to 30 months); based on cutoff date: 19 September 2018.
Population: The primary analyses of PFS based on BICR assessment were performed using FAS. The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
months | 1.9 [1.8 to 1.9] | 3.7 [3.3 to 5.1] | 3.5 [2.1 to 4.0]
Statistical Analysis 1: Comparison: Avelumab vs Pegylated Liposomal Doxorubicin (PLD); Test type: Superiority; p > 0.9999, Log Rank; 1-sided; Hazard Ratio (HR) = 1.68, 95% CI 2-sided [1.310 to 2.160]
Statistical Analysis 2: Comparison: Avelumab + PLD vs Pegylated Liposomal Doxorubicin (PLD); Test type: Superiority; p = 0.0301, Log Rank; 1-sided; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.607 to 1.011]

3. Secondary Outcome: Objective Response Rate (ORR) Based on BICR Assessment
Description: Percentage of participants achieved objective response (OR) based on BICR assessment is presented for this endpoint. OR is defined as a complete response (CR, disappearance of all target lesions) or partial response (PR, >=30% decrease under the baseline of the sum of diameters of all target measurable lesions) according to the RECIST (version 1.1) recorded from randomization until disease progression or death due to any cause. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met and before the first documentation of disease progression. Only tumor assessments performed on or before the start date of any further anti-cancer therapies are considered in the assessment of best overall response.
Time Frame: Tumor assessments as assessed by BICR were conducted at every 8 weeks from screening until documented disease progression (approximately up to 30 months); based on cutoff date: 19 September 2018.
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
percentage of participants | 3.7 [1.5 to 7.5] | 13.3 [8.8 to 19.0] | 4.2 [1.8 to 8.1]

4. Secondary Outcome: ORR Based on Investigator Assessment
Description: Percentage of participants achieved OR based on investigator assessment is presented for this endpoint. OR is defined as a CR (disappearance of all target lesions) or PR (>=30% decrease under the baseline of the sum of diameters of all target measurable lesions) according to the RECIST (version 1.1) recorded from randomization until disease progression or death due to any cause. The ORR on each randomized treatment arm were estimated by dividing the number of participants with OR (CR or PR) by number of participants randomized to the respective treatment arm.
Time Frame: Tumor assessments as assessed by investigator were conducted at every 8 weeks from screening until documented disease progression, up to 30 months; based on cutoff date: 19 September 2018.
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
percentage of participants | 5.3 [2.6 to 9.6] | 18.6 [13.3 to 24.9] | 9.5 [5.7 to 14.6]

5. Secondary Outcome: PFS Based on Investigator Assessment According to RECIST Version 1.1
Description: PFS is defined as the time from date of randomization to the date of the first documentation of PD or death due to any cause, whichever occurs first. PFS time was summarized by treatment arm using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
month | 1.9 [1.8 to 1.9] | 4.7 [3.7 to 6.0] | 3.7 [3.5 to 5.4]

6. Secondary Outcome: Duration of Response (DR) Based on BICR Assessment
Description: DR is defined, for participants with an OR per RECIST version 1.1, as the time from the first documentation of objective tumor response (CR [disappearance of all target lesions] or PR [>=30% decrease under the baseline of the sum of diameters of all target measurable lesions]) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first.
Time Frame: as for outcome 4
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were randomized. Number analyzed are participants with confirmed CR or PR in the FAS within each treatment group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 7 | 25 | 8
months | 9.2 [6.4 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to the small number of events. | 8.5 [6.1 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 13.1 [5.5 to NA] — The upper limit of 95% CI was not estimable due to the small number of events.

7. Secondary Outcome: DR Based on Investigator Assessment
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 10 | 35 | 18
months | 10.4 [3.7 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 7.6 [5.6 to 9.1] | 7.4 [3.6 to 11.2]

8. Secondary Outcome: Disease Control (DC) Rate Based on BICR Assessment
Description: Percentage of participants achieving DC based on BICR assessment is presented in this endpoint. DC is a best overall response of CR (disappearance of all target lesions), PR (>=30% decrease under the baseline of the sum of diameters of all target measurable lesions), non-complete response/non-progressive disease or stable disease (SD) according to the RECIST version 1.1.
Time Frame: as for outcome 4
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
percentage of participants | 33.0 [26.3 to 40.2] | 57.4 [50.0 to 64.6] | 48.9 [41.6 to 56.3]

9. Secondary Outcome: DC Rate Based on Investigator Assessment
Description: Percentage of participants achieving DC based on investigator assessment is presented in this endpoint. DC is a best overall response of CR (disappearance of all target lesions), PR (>=30% decrease under the baseline of the sum of diameters of all target measurable lesions), non-complete response/non-progressive disease or SD according to the RECIST version 1.1.
Time Frame: as for outcome 4
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
percentage of participants | 34.0 [27.3 to 41.3] | 61.7 [54.3 to 68.7] | 54.7 [47.4 to 62.0]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; progression of the malignancy under study. Treatment emergent AEs are those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event is during the on-treatment period.
Time Frame: From the time of the first dose of study treatment through a minimum of 30 days + last dose of study treatment, start day of new anti-cancer therapy -1 day (up to 70 months); based on cutoff date: 13 July 2022.
Population: Analysis is based on the safety analysis set. The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 187 | 182 | 177
Participants
  TEAE | 180 | 180 | 173
  Treatment emergent SAEs | 72 | 74 | 51

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: The number of participants with following laboratory abnormalities meeting any of the Grades 1 to 4 classified according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading version 4.03 were summarized: hematology (anemia, lymphocyte count decreased, neutrophil count decreased; and platelet count decreased) and chemistry laboratory tests (creatinine increased; serum amylase increased and lipase increased).
Time Frame: From screening to the end of treatment/withdrawal visit, up to 2.7 years, based on cutoff date: 19 September 2018.
Population: 'Number of Participants Analyzed' is based on the safety analysis set, which included all participants who received at least 1 dose of study treatment. 'Number Analyzed' included the number of participants in the safety analysis set who can be evaluated for CTCAE criteria for each parameter in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 187 | 182 | 177
Participants
  Anemia: number analyzed (Participants) | 186 | 178 | 172
  Anemia | 135 | 155 | 144
  Lymphocyte count decreased: number analyzed (Participants) | 185 | 178 | 171
  Lymphocyte count decreased | 89 | 148 | 107
  Neutrophil count decreased: number analyzed (Participants) | 185 | 177 | 172
  Neutrophil count decreased | 26 | 80 | 62
  Platelet count decreased: number analyzed (Participants) | 186 | 178 | 172
  Platelet count decreased | 33 | 48 | 50
  Creatinine increased: number analyzed (Participants) | 186 | 178 | 172
  Creatinine increased | 154 | 151 | 120
  Serum amylase increased: number analyzed (Participants) | 180 | 172 | 161
  Serum amylase increased | 43 | 35 | 27
  Lipase increased: number analyzed (Participants) | 175 | 173 | 159
  Lipase increased | 27 | 33 | 21

12. Secondary Outcome: Change From Baseline in Vital Signs - Blood Pressure
Description: Vital signs included blood pressure and pulse rate. Changes from baseline in sitting diastolic blood pressure (DBP) and systolic blood pressure (SBP) were summarized.
Time Frame: From screening to the end of treatment/withdrawal visit, up to 2.7 years, based on cutoff date: 19 September 2018.
Population: 'Number of Participants Analyzed' is based on the safety analysis set, which included all participants who received at least 1 dose of study treatment. 'Number Analyzed' included the number of participants in the safety analysis set with at least a baseline and post-baseline assessment at the visit.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 187 | 182 | 177
mm Hg
  DBP Cycle 1 Day 15: number analyzed (Participants) | 180 | 170 | 142
  DBP Cycle 1 Day 15 | 0.1 (9.79) | -2.2 (9.12) | 0.7 (8.89)
  DBP Cycle 2 Day 1: number analyzed (Participants) | 164 | 168 | 156
  DBP Cycle 2 Day 1 | -1.1 (9.61) | -2.8 (8.01) | -0.1 (9.34)
  DBP Cycle 2 Day 15: number analyzed (Participants) | 138 | 157 | 124
  DBP Cycle 2 Day 15 | 0.1 (10.05) | -2.8 (9.19) | -0.1 (8.83)
  DBP Cycle 3 Day 1: number analyzed (Participants) | 104 | 141 | 106
  DBP Cycle 3 Day 1 | 0 (10.81) | -2.7 (8.95) | -0.2 (8.96)
  DBP Cycle 3 Day 15: number analyzed (Participants) | 95 | 128 | 84
  DBP Cycle 3 Day 15 | -0.6 (9.25) | -2.3 (8.56) | -0.5 (8.67)
  DBP End of Treatment: number analyzed (Participants) | 146 | 138 | 136
  DBP End of Treatment | 1.1 (10.87) | -0.3 (11.08) | 0.8 (10.40)
  SBP Cycle 1 Day 15: number analyzed (Participants) | 180 | 170 | 142
  SBP Cycle 1 Day 15 | -0.9 (14.35) | -2.3 (13.12) | -1.0 (13.94)
  SBP Cycle 2 Day 1: number analyzed (Participants) | 164 | 168 | 156
  SBP Cycle 2 Day 1 | -2.2 (14.44) | -3.4 (13.70) | -2.8 (13.39)
  SBP Cycle 2 Day 15: number analyzed (Participants) | 138 | 157 | 124
  SBP Cycle 2 Day 15 | -0.6 (14.11) | -3.7 (14.78) | -1.8 (14.98)
  SBP Cycle 3 Day 1: number analyzed (Participants) | 104 | 141 | 106
  SBP Cycle 3 Day 1 | -0.2 (15.59) | -2.7 (14.36) | -1.5 (14.14)
  SBP Cycle 3 Day 15: number analyzed (Participants) | 95 | 128 | 84
  SBP Cycle 3 Day 15 | -0.2 (13.78) | -2.1 (15.30) | -2.2 (13.96)
  SBP End of Treatment: number analyzed (Participants) | 146 | 138 | 136
  SBP End of Treatment | -0.9 (17.21) | -1.0 (16.83) | -3.2 (15.92)

13. Secondary Outcome: Change From Baseline in Vital Signs - Pulse Rate
Description: Vital signs included blood pressure and pulse rate. Changes from baseline in sitting pulse rate were summarized.
Time Frame: From screening to the end of treatment/withdrawal visit, up to 2.7 years, based on cutoff date: 19 September 2018.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 187 | 182 | 177
bpm
  Cycle 1 Day 15: number analyzed (Participants) | 180 | 170 | 142
  Cycle 1 Day 15 | 2.9 (9.95) | 1.8 (12.10) | 3.5 (10.70)
  Cycle 2 Day 1: number analyzed (Participants) | 164 | 167 | 155
  Cycle 2 Day 1 | 2.6 (10.92) | 2.9 (11.18) | 1.7 (9.71)
  Cycle 2 Day 15: number analyzed (Participants) | 138 | 157 | 124
  Cycle 2 Day 15 | 2.9 (11.19) | 3.5 (11.79) | 3.2 (11.54)
  Cycle 3 Day 1: number analyzed (Participants) | 104 | 141 | 106
  Cycle 3 Day 1 | 2.4 (10.00) | 2.1 (11.78) | 1.4 (11.14)
  Cycle 3 Day 15: number analyzed (Participants) | 95 | 128 | 84
  Cycle 3 Day 15 | 3.0 (12.23) | 1.4 (11.44) | 2.4 (10.41)
  End of Treatment: number analyzed (Participants) | 146 | 138 | 136
  End of Treatment | 7.7 (14.27) | 7.4 (13.70) | 5.7 (14.10)

14. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Categorical summarization ECG criteria were as follows: 1) QT interval, QTcB, QTcF and QTcP: increase from baseline >30 ms or 60 ms; absolute value > 450 ms, >480 ms and > 500 ms; 2) heart rate (HR): change from baseline >=20 bpm and absolute value <=50 bpm or >=120 bpm; 3) PR interval: absolute value >=220 ms and increase from baseline >=20 ms; 4) QRS: >= 120 ms.
Time Frame: From screening to the end of treatment/withdrawal visit, up to 2.7 years, based on cutoff date: 19 September 2018.
Population: 'Number of Participants Analyzed' is based on the safety analysis set, which included all participants who received at least 1 dose of study treatment. 'Number Analyzed' included the number of participants in the safety analysis set who had a at least 1 post-baseline ECG assessment performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 187 | 182 | 177
Participants
  QT increase from baseline >30 ms: number analyzed (Participants) | 183 | 176 | 169
  QT increase from baseline >30 ms | 26 | 40 | 47
  QT increase from baseline >60 ms: number analyzed (Participants) | 183 | 176 | 169
  QT increase from baseline >60 ms | 5 | 9 | 4
  QT >450 ms: number analyzed (Participants) | 183 | 176 | 169
  QT >450 ms | 6 | 10 | 5
  QT >480 ms: number analyzed (Participants) | 183 | 176 | 169
  QT >480 ms | 1 | 2 | 2
  QT >500 ms: number analyzed (Participants) | 183 | 176 | 169
  QT >500 ms | 1 | 1 | 1
  QTcB increase from baseline >30 ms: number analyzed (Participants) | 154 | 153 | 143
  QTcB increase from baseline >30 ms | 33 | 36 | 22
  QTcB increase from baseline >60 ms: number analyzed (Participants) | 154 | 153 | 143
  QTcB increase from baseline >60 ms | 9 | 7 | 8
  QTcB >450 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcB >450 ms | 56 | 63 | 45
  QTcB >480 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcB >480 ms | 9 | 19 | 9
  QTcB >500 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcB >500 ms | 5 | 9 | 5
  QTcF increase from baseline >30 ms: number analyzed (Participants) | 154 | 153 | 143
  QTcF increase from baseline >30 ms | 19 | 24 | 13
  QTcF increase from baseline >60 ms: number analyzed (Participants) | 154 | 153 | 143
  QTcF increase from baseline >60 ms | 6 | 5 | 5
  QTcF >450 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcF >450 ms | 18 | 27 | 14
  QTcF >480 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcF >480 ms | 4 | 8 | 5
  QTcF >500 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcF >500 ms | 3 | 2 | 4
  QTcP increase from baseline >30 ms: number analyzed (Participants) | 154 | 153 | 143
  QTcP increase from baseline >30 ms | 17 | 23 | 12
  QTcP increase from baseline >60 ms: number analyzed (Participants) | 154 | 153 | 143
  QTcP increase from baseline >60 ms | 6 | 5 | 4
  QTcP >450 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcP >450 ms | 19 | 29 | 17
  QTcP >480 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcP >480 ms | 2 | 7 | 2
  QTcP >500 ms: number analyzed (Participants) | 161 | 160 | 145
  QTcP >500 ms | 1 | 2 | 2
  Heart rate <=50 bpm and decrease >= 20 bpm: number analyzed (Participants) | 154 | 153 | 143
  Heart rate <=50 bpm and decrease >= 20 bpm | 0 | 1 | 0
  Heart rate >=120 bpm and increase >= 20 bpm: number analyzed (Participants) | 154 | 153 | 143
  Heart rate >=120 bpm and increase >= 20 bpm | 5 | 5 | 3
  PR >=220 ms and increase from baseline >=20 ms: number analyzed (Participants) | 182 | 176 | 168
  PR >=220 ms and increase from baseline >=20 ms | 3 | 4 | 2
  QRS >=120 ms: number analyzed (Participants) | 183 | 176 | 169
  QRS >=120 ms | 7 | 9 | 9

15. Secondary Outcome: Number of Participants With % Left Ventricular Ejection Fraction (LVEF) Decrease From Baseline
Description: LVEF decrease was summarized by multiple-gated acquisition (MUGA)/ echocardiogram (ECHO) parameter. Participants with a LVEF% >=10 points and >= 15 points decrease from baseline during the on-treatment period were summarized.
Time Frame: Screening, Cycle 3 Day 1 (repeated every 2 cycles) to the end of treatment/withdrawal visit, based on cutoff date: 19 September 2018.
Population: 'Number of Participants Analyzed' is based on number of participants in the safety analysis set with a baseline and a post-baseline assessment within each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 129 | 154 | 132
Participants
  >= 10 point decrease from baseline | 8 | 22 | 13
  >= 15 point decrease from baseline | 3 | 8 | 3

16. Secondary Outcome: Number of Participants With PD-L1 Expression for PFS (Based on BICR Assessment) and for OS
Description: PD-L1 expression was assessed by immunohistochemistry. Participants were considered positive for PD-L1 if their baseline tissue sample demonstrated PD-L1 expression on >=1% of tumor cells or >=5% of immune cells.
Time Frame: Biomarkers are measured only at screening.
Population: The biomarker analysis set included participants who had at least 1 screening biomarker assessment. 'Number of Participants Analyzed' is based on number of participants in the biomarker analysis set within each treatment group with reported PD-L1 status.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 170 | 173 | 165
Participants | 100 | 100 | 88

17. Secondary Outcome: Number of Participants With CD8 Expression for PFS (Based on BICR Assessment) and for OS
Description: Tumor infiltrating CD8 positive (CD8+) T lymphocytes was assessed by immunohistochemistry. Participants were considered positive for CD8 T cells if their baseline tissue sample demonstrated presence of >=1% CD8+ cells across the area of the tumor.
Time Frame: Biomarkers are measured only at screening.
Population: The biomarker analysis set included participants who had at least 1 screening biomarker assessment. 'Number of Participants Analyzed' is based on number of participants in the biomarker analysis set within each treatment group with reported CD8 status.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 165 | 171 | 164
Participants | 76 | 80 | 72

18. Secondary Outcome: Number of Participants With Improved, Stable and Deterioration Based on 10-Point Change for EORTC QLQ-C30 Global QoL
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) is a 30 question survey and includes 5 functional domain subscales, global health status/quality of life, disease/treatment related symptoms, and the perceived financial impact of disease. Higher scores are reflective of a greater presence of symptoms.
Time Frame: Day 1 of Cycle 1, Day 1 of each subsequent cycle, end of treatment/withdrawal visit and the 30, 60 and 90 days safety follow up visits, based on cutoff date: 19 September 2018.
Population: The analysis is based on the FAS. The FAS included all participants who were randomized. 'Number Analyzed' in represents number of participants in the FAS with a score at baseline and post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 152 | 166 | 148
Participants
  Deterioration | 46 | 65 | 46
  Improved | 23 | 20 | 26
  Stable | 83 | 81 | 76

19. Secondary Outcome: Time to Deterioration in Abdominal/GI Symptom Subscale of EORTC QLQ-OV28
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Ovarian Cancer 28 (EORTC QLQ-OV28) is a 28 item instrument with 7 functional domain subscales. Time to deterioration was defined as the time from randomization to the first time the participant's score showed a 15-point or higher increase in the score of the abdominal/GI symptom subscale of the EORTC QLQ-OV28.
Time Frame: From Day 1 of Cycle 1 to prior to end of treatment/withdrawal visit, based on cutoff date: 19 September 2018.
Population: The analysis is based on the FAS. The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 188 | 188 | 190
months | NA [NA to NA] — The median estimates of time to event, upper and lower limits of 95% CI were not estimable due to the small number of events. | 11.1 [6.5 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 10.6 [9.2 to NA] — The upper limit of 95% CI was not estimable due to the small number of events.

20. Secondary Outcome: Change From Baseline in EQ-VAS Score at End of Treatment
Description: The EuroQol- 5 Dimensions- 5 Levels (EQ-5D-5L) questionnaire consists of the EQ-5D-5L descriptive system and a visual analogue scale (the EuroQol-visual analogue scale [EQ-VAS]). The respondent's self-rated health is assessed on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state) by the EQ-VAS.
Time Frame: Baseline and end of treatment/withdrawal visit
Population: The analysis is based on the FAS. The FAS included all participants who were randomized. 'Number Analyzed' represents number of participants in the FAS with an assessment at the visit or with at least a baseline and post-baseline assessment at visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
Number analyzed (Participants) | 111 | 116 | 111
scores on a scale | -13.6 (20.56) | -11.2 (19.79) | -7.7 (22.26)

21. Secondary Outcome: Serum Trough Concentration (Ctrough) For Avelumab Following Cycle 2 Day 1 Pegylated Liposomal Doxorubicin (PLD) Dose
Description: Ctrough was defined as predose concentration during multiple dosing, and can be observed directly from data.
Time Frame: At predose (0 H) on Cycle 2 Day 1
Population: The PK parameter analysis set was defined as participants in the safety analysis set who had at least 1 post-dose concentration measurement above the lower limit of quantitation (LLQ) for avelumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Avelumab | Avelumab + PLD
Number analyzed (Participants) | 136 | 139
microgram per milliliter (mcg/mL) | 21.1 (89) | 23.19 (74)
Statistical Analysis 1: Comparison: Avelumab vs Avelumab + PLD; Avelumab was the Reference treatment and Avelumab + PLD was the Test treatment; Test type: Other; Geometric Mean Ratio (Test/Reference, %) = 110, 90% CI 2-sided [95.4 to 126.7]

22. Secondary Outcome: Serum Maximum Concentration (Cmax) For Avelumab Following Cycle 2 Day 1 PLD Dose
Description: Cmax was defined as maximum observed serum concentration, and can be observed directly from data.
Time Frame: At postdose (end of infusion, 1H) on Cycle 2 Day 1
Population: The PK parameter analysis set was defined as participants in the safety analysis set who had at least 1 post-dose concentration measurement above the LLQ for avelumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Avelumab | Avelumab + PLD
Number analyzed (Participants) | 104 | 110
mcg/mL | 231.6 (43) | 207.9 (71)
Statistical Analysis 1: Comparison: Avelumab vs Avelumab + PLD; Avelumab was the Reference treatment and Avelumab + PLD was the Test treatment; Test type: Other; Geometric Mean Ratio (Test/Reference, %) = 90, 90% CI 2-sided [79.5 to 101.5]

23. Secondary Outcome: Cmax For Doxorubicin Following Cycle 2 Day 1 PLD Dose
Description: Cmax was defined as maximum observed serum concentration, and can be observed directly from data.
Time Frame: From predose (0 H) of Cycle 2 Day 1 through 336 hours postdose
Population: The PK parameter analysis set was defined as a subset of the safety analysis set and included patients who had at least one of the PK parameters of interest for doxorubicin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Avelumab + PLD
Number analyzed (Participants) | 15 | 15
nanogram per milliliter (ng/mL) | 26810 (14) | 25850 (17)
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Avelumab + PLD; PLD was the Reference treatment and Avelumab + PLD was the Test treatment; Test type: Other; Geometric Mean Ratio (Test/Reference, %) = 96, 90% CI 2-sided [87 to 106]

24. Secondary Outcome: Area Under The Concentration Time Profile From Time Zero to 24 Hours (AUC24) For Doxorubicin Following Cycle 2 Day 1 PLD Dose
Description: AUC24 was defined as area under the concentration time profile from time zero to 24 hours.
Time Frame: From 0 through 24 hours postdose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Avelumab + PLD
Number analyzed (Participants) | 14 | 14
nanogram*hour per milliliter (ng*hr/mL) | 567600 (11) | 541700 (14)
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Avelumab + PLD; PLD was the Reference treatment and Avelumab + PLD was the Test treatment; Test type: Other; Geometric Mean Ratio (Test/Reference, %) = 95, 90% CI 2-sided [88 to 104]

25. Secondary Outcome: Area Under The Concentration Time Profile From Time Zero to 336 Hours (AUC336) For Doxorubicin Following Cycle 2 Day 1 PLD Dose
Description: AUC336 was defined as area under the concentration time profile from time zero to 336 hours.
Time Frame: From predose (0 H) of Cycle 2 Day 1 through 336 hours postdose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Avelumab + PLD
Number analyzed (Participants) | 13 | 12
ng*hr/mL | 2848000 (20) | 2571000 (30)
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Avelumab + PLD; PLD was the Reference treatment and Avelumab + PLD was the Test treatment; Test type: Other; Geometric Mean Ratio (Test/Reference, %) = 90, 90% CI 2-sided [76 to 107]

26. Secondary Outcome: Area Under The Concentration Time Profile From Time Zero to The Last Quantifiable Concentration (AUClast) For Doxorubicin Following Cycle 2 Day 1 PLD Dose
Description: AUClast was defined as area under the concentration time profile from time zero to the time of the last quantifiable concentration (Clast).
Time Frame: From predose (0 H) of Cycle 2 Day 1 through 336 hours postdose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) | Avelumab + PLD
Number analyzed (Participants) | 15 | 15
ng*hr/mL | 2043000 (119) | 2052000 (71)
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) vs Avelumab + PLD; PLD was the Reference treatment and Avelumab + PLD was the Test treatment; Test type: Other; Geometric Mean Ratio (Test/Reference, %) = 100, 90% CI 2-sided [60 to 168]

27. Secondary Outcome: Number of Participants With Treatment-Boosted Anti-Drug Antibody (ADA)
Description: Treatment-boosted ADA was defined as a positive ADA result at baseline and the titer ≥ 8×baseline titer at least once after treatment with avelumab.
Time Frame: At predose (0 H) of select cycles starting from Cycle 1 through Cycle 24, at end of treatment and 30 days after the last dose of avelumab
Population: The analysis set was defined as participants with valid baseline ADA results and at least one valid post-baseline ADA result in the immunogenicity analysis set. The immunogenicity analysis set was a subset of the safety analysis set and included patients who had at least one ADA/nAb sample collected for avelumab in the avelumab containing arms.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Total participants from the 2 arms.
Arm/Group | Avelumab | Avelumab + PLD | All Participants
Number analyzed (Participants) | 165 | 167 | 332
Participants | 1 | 0 | 1

28. Secondary Outcome: Number of Participants With Treatment-Induced ADA
Description: Treatment-induced ADA was defined as participant who was ADA-negative at baseline and has at least one positive post-baseline ADA result; or if participant did not have a baseline sample, the participant had at least one positive past-baseline ADA result.
Time Frame: as for outcome 27
Population: The analysis set was defined as participants with at least 1 valid post-baseline ADA results and without positive baseline ADA result in the immunogenicity analysis set. The immunogenicity analysis set was a subset of the safety analysis set and included patients who had at least one ADA/nAb sample collected for avelumab in the avelumab containing arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | All Participants
Number analyzed (Participants) | 169 | 167 | 336
Participants | 27 | 2 | 29

29. Secondary Outcome: Number of Participants With Treatment-Induced Neutralizing Antibody (nAb)
Description: Treatment-induced nAb was defined as participant who was not nAb positive at baseline and had at least one positive post-baseline nAb result; or if participant did not have a baseline sample, the participant had at least one positive past-baseline ADA result.
Time Frame: as for outcome 27
Population: The analysis set was defined as participants with at least 1 valid post-baseline ADA result and without positive baseline nAb result in the immunogenicity analysis set. The immunogenicity analysis set was a subset of the safety analysis set and included patients who had at least one ADA/nAb sample collected for avelumab in the avelumab containing arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Avelumab + PLD | All Participants
Number analyzed (Participants) | 173 | 169 | 342
Participants | 5 | 1 | 6

ADVERSE EVENTS:
Time Frame: AEs (serious and non-serious) should be reported from the time of the first dose of study treatment through a minimum of 30 days + last dose of study treatment, start day of new anti-cancer therapy -1 day (up to 70 months). Based on the cutoff: 13 July 2022.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. The mortality analysis set included all randomized participants. The AE and SAE analysis set included participants who received at least 1 dose of study drug.
Arm/Group | Avelumab | Avelumab + PLD | Pegylated Liposomal Doxorubicin (PLD)
All-Cause Mortality (participants affected / at risk) | 122/187 | 107/182 | 116/177
Serious Adverse Events (participants affected / at risk) | 72/187 | 74/182 | 51/177
Other Adverse Events (participants affected / at risk) | 173/187 | 176/182 | 167/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=187) | Avelumab + PLD (N=182) | Pegylated Liposomal Doxorubicin (PLD) (N=177)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 10 (10) | 5 (5) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 8 (9) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 6 (6) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (3) | 1 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 11 (16) | 9 (9) | 6 (6)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 4 (4) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8) | 4 (4) | 3 (5)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated adverse reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Septic pulmonary embolism (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Clonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=187) | Avelumab + PLD (N=182) | Pegylated Liposomal Doxorubicin (PLD) (N=177)
Anaemia (Blood and lymphatic system disorders) | 32 (68) | 56 (131) | 42 (77)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 27 (58) | 25 (52)
Hypothyroidism (Endocrine disorders) | 9 (11) | 20 (22) | 2 (2)
Asthenia (General disorders) | 18 (27) | 30 (68) | 14 (18)
Chills (General disorders) | 18 (20) | 14 (15) | 3 (3)
Fatigue (General disorders) | 63 (88) | 77 (147) | 55 (78)
Influenza like illness (General disorders) | 6 (7) | 10 (13) | 1 (1)
Malaise (General disorders) | 5 (5) | 11 (14) | 6 (6)
Mucosal inflammation (General disorders) | 4 (7) | 24 (45) | 19 (29)
Oedema peripheral (General disorders) | 13 (16) | 24 (32) | 14 (16)
Pyrexia (General disorders) | 27 (32) | 36 (61) | 16 (20)
Abdominal distension (Gastrointestinal disorders) | 14 (19) | 18 (21) | 18 (20)
Abdominal pain (Gastrointestinal disorders) | 54 (69) | 47 (67) | 38 (48)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 17 (22) | 13 (13)
Ascites (Gastrointestinal disorders) | 12 (16) | 5 (9) | 4 (7)
Constipation (Gastrointestinal disorders) | 35 (47) | 48 (69) | 46 (58)
Diarrhoea (Gastrointestinal disorders) | 42 (61) | 36 (57) | 32 (45)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 18 (25) | 14 (15)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (9) | 9 (11) | 14 (17)
Nausea (Gastrointestinal disorders) | 53 (66) | 87 (131) | 76 (117)
Stomatitis (Gastrointestinal disorders) | 8 (13) | 53 (125) | 35 (73)
Vomiting (Gastrointestinal disorders) | 43 (63) | 43 (65) | 44 (58)
Urinary tract infection (Infections and infestations) | 15 (22) | 20 (29) | 12 (21)
Infusion related reaction (Injury, poisoning and procedural complications) | 13 (17) | 17 (20) | 14 (14)
Alanine aminotransferase increased (Investigations) | 4 (8) | 16 (22) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 4 (7) | 18 (30) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 11 (20) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 13 (16) | 13 (30) | 6 (9)
Lymphocyte count decreased (Investigations) | 1 (1) | 13 (54) | 4 (4)
Neutrophil count decreased (Investigations) | 4 (10) | 17 (84) | 9 (33)
Platelet count decreased (Investigations) | 5 (8) | 10 (22) | 7 (16)
Weight decreased (Investigations) | 10 (11) | 13 (19) | 13 (19)
White blood cell count decreased (Investigations) | 6 (7) | 15 (70) | 15 (41)
Decreased appetite (Metabolism and nutrition disorders) | 36 (41) | 51 (69) | 37 (45)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (16) | 13 (24) | 6 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (12) | 12 (17) | 11 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (12) | 8 (15) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (22) | 17 (20) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (25) | 18 (28) | 21 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 14 (21) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 18 (20) | 13 (14)
Dizziness (Nervous system disorders) | 5 (5) | 17 (19) | 8 (8)
Headache (Nervous system disorders) | 15 (16) | 29 (34) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 28 (45) | 24 (27)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (45) | 32 (44) | 25 (32)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (12) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 18 (18) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 23 (25) | 8 (9)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 61 (163) | 40 (74)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (14) | 21 (34) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 12 (21) | 51 (126) | 21 (26)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 14 (40) | 11 (19)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (10) | 10 (10)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 10 (12) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (15) | 5 (7)
Anxiety (Psychiatric disorders) | 7 (7) | 10 (11) | 6 (7)
C-reactive protein increased (Investigations) | 0 (0) | 10 (13) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02580058/Prot_002.pdf
  • Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02580058/SAP_000.pdf